CLINICAL TRIAL: NCT07395375
Title: A Multicenter, Randomized, Controlled Trial of Non-Intubated Spontaneous Breathing Anesthesia Versus Intubated Mechanical Ventilation Anesthesia in Thoracoscopic Sublobar Resection: A Stratified Analysis Study Focusing on Safety and Recovery Quality
Brief Title: Non-intubated Versus Intubated Anesthesia for Thoracoscopic Sublobar Resection
Acronym: NIVA-TSLR
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: The First Affiliated Hospital of Guangzhou Medical University (Other)
Responsible Party: Principal Investigator, Jianxing He, Professor, Chief of Thoracic Surgery Department, The First Affiliated Hospital of Guangzhou Medical University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: NIT-Sublobar-VATS
Record Dates: First submitted 2026-01-24; First posted 2026-02-09 (Actual); Last update posted 2026-02-09 (Actual); Status verified 2026-01

CONDITIONS: Pulmonary Nodules; Lung Neoplasms; Thoracic Surgery
Keywords: Non-intubated Thoracic Surgery; Lung Sublobar Resection; Video-Assisted Thoracoscopic Surgery; Enhanced Recovery After Surgery; Randomized Controlled Trial
MeSH Terms: conditions — Multiple Pulmonary Nodules; Lung Neoplasms | interventions — Laryngeal Masks; Anesthesia; Anesthesia, General; Neuromuscular Blockade

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Non-intubated Anesthesia Group (Experimental): Patients randomized to this group will receive the experimental intervention, non-intubated spontaneous breathing anesthesia. The key components include:
  Airway Management: A laryngeal mask airway will be used instead of an endotracheal tube.
  Anesthesia Technique: Intravenous sedation will be administered to maintain spontaneous breathing, combined with regional nerve blocks (e.g., paravertebral or intercostal block) for analgesia.
  Goal: This approach aims to avoid the potential trauma and lung injury associated with double-lumen tube intubation and mechanical ventilation.
  A predefined set of safety criteria for conversion to intubated anesthesia (e.g., low oxygen levels, excessive carbon dioxide buildup) will be strictly followed during the procedure.
  Interventions: Procedure: Non-intubated Anesthesia; Device: Laryngeal Mask Airway (LMA); Drug: Intravenous Sedation/Anesthesia (Spontaneous Ventilation); Drug: Regional Nerve Block (Paravertebral/Intercostal Block)
- Conventional Anesthesia Group (Active Comparator): Patients randomized to this group will receive the current standard of care for thoracoscopic lung surgery, which is conventional intubated general anesthesia. The intervention consists of:
  Airway Management: Double-lumen endobronchial tube intubation to achieve one-lung ventilation.
  Anesthesia Technique: Standard general anesthesia with muscle relaxation and controlled mechanical ventilation.
  This approach represents the well-established, traditional method against which the experimental non-intubated anesthesia is being compared.
  Interventions: Procedure: Conventional Intubated General Anesthesia; Device: Double-lumen Endotracheal Tube (DLT); Drug: General Anesthesia With Neuromuscular Blockade

INTERVENTIONS:
Procedure: Non-intubated Anesthesia — A novel anesthetic technique for thoracic surgery that avoids endotracheal intubation and mechanical ventilation. It typically involves intravenous sedation, the use of a laryngeal mask airway (LMA) for oxygenation, and regional nerve blocks (e.g., paravertebral block) for pain control. The key feature is the preservation of the patient's spontaneous breathing throughout the surgical procedure.
  Arms: Non-intubated Anesthesia Group
Procedure: Conventional Intubated General Anesthesia — The current standard anesthetic technique for thoracoscopic surgery. It involves general anesthesia induced by intravenous agents, followed by the insertion of a double-lumen endotracheal tube to achieve one-lung ventilation. Anesthesia is maintained with inhalational or intravenous agents, and the patient's ventilation is fully controlled by a mechanical ventilator throughout the operation.
  Arms: Conventional Anesthesia Group
Device: Laryngeal Mask Airway (LMA) — Airway management using a laryngeal mask airway to maintain spontaneous ventilation during thoracoscopic surgery.
  Arms: Non-intubated Anesthesia Group
Drug: Intravenous Sedation/Anesthesia (Spontaneous Ventilation) — Intravenous sedative/anesthetic agents administered to achieve adequate anesthesia while preserving spontaneous breathing.
  Arms: Non-intubated Anesthesia Group
Drug: Regional Nerve Block (Paravertebral/Intercostal Block) — Regional anesthesia with local anesthetic (e.g., paravertebral or intercostal block) for perioperative analgesia.
  Arms: Non-intubated Anesthesia Group
Device: Double-lumen Endotracheal Tube (DLT) — Double-lumen endotracheal tube used to achieve one-lung ventilation during general anesthesia.
  Arms: Conventional Anesthesia Group
Drug: General Anesthesia With Neuromuscular Blockade — General anesthesia maintained with intravenous and/or inhalational agents with muscle relaxation for controlled mechanical ventilation.
  Arms: Conventional Anesthesia Group

SUMMARY:
This is a large clinical study that compares two different types of anesthesia for patients undergoing a specific kind of minimally invasive lung surgery (thoracoscopic sublobar resection) to remove small, early-stage lung nodules.

The study aims to find out if a newer anesthesia method, known as "non-intubated anesthesia" (where patients breathe on their own with the help of a laryngeal mask airway and nerve blocks for pain control), is as safe as the traditional "intubated anesthesia" (which uses a breathing tube and a machine to breathe for the patient).

The main goals of the study are, in order:

1. Safety First: To confirm that the non-intubated method does not lead to more lung complications within 30 days after surgery compared to the traditional method.
2. Effectiveness: If it is proven safe, the study will then check if patients receiving the non-intubated anesthesia have a better quality of recovery in the first 24 hours after surgery (e.g., less pain, fewer side effects like a sore throat, and a faster return to normal activities).

Approximately 1600 patients from multiple hospitals will be randomly assigned (like flipping a coin) to receive one of the two anesthesia methods. Neither the patients nor the surgeons will be told which group the patient is in when assessing the main outcomes after surgery, to ensure the results are fair and unbiased.

The results of this study will provide high-quality evidence to help doctors and patients choose the best and most comfortable anesthesia option for this type of lung surgery.

ELIGIBILITY:
Inclusion Criteria:

1. Aged 18 to 80 years (inclusive).
2. Scheduled for elective, uniportal or single utility port video-assisted thoracoscopic sublobar resection (wedge resection or simple anatomical segmentectomy).
3. Preoperative CT diagnosis of a peripheral pulmonary nodule meeting: maximum diameter ≤ 2.0 cm and outer edge ≤ 2.0 cm from the visceral pleura.
4. American Society of Anesthesiologists (ASA) physical status I or II.
5. Preoperative pulmonary function: FEV1% ≥ 60% of predicted.
6. Preoperative arterial blood gas analysis (room air): PaO₂ ≥ 80 mmHg and PaCO₂ ≤ 45 mmHg.
7. Body Mass Index (BMI) between 18.0 and 28.0 kg/m².
8. Able to understand the study and provide written informed consent.

Exclusion Criteria:

1. Cardiovascular: NYHA class ≥ III, unstable angina, acute myocardial infarction within 3 months, or severe arrhythmia requiring medication.
2. Respiratory: Severe COPD (GOLD 3 or 4), symptomatic interstitial lung disease, resting SpO₂ < 92% on room air, or severe pulmonary hypertension (estimated systolic PAP > 50 mmHg).
3. Airway Risk: Modified Mallampati score ≥ 3, mouth opening < 3 cm, or other predictors of difficult airway management.
4. Radiological: Preoperative CT suggesting extensive pleural adhesion, moderate or large pleural effusion, or mediastinal lymph nodes > 1.5 cm short axis.
5. Contraindications to Regional Anesthesia: Infection/tumor at the block site, patient refusal, or allergy to local anesthetics.
6. Coagulopathy: Platelet count < 100×10⁹/L, INR > 1.5, or use of anticoagulants that cannot be safely discontinued perioperatively.
7. Other: Severe hepatic or renal dysfunction, previous ipsilateral thoracic surgery, pregnancy or lactation, active psychiatric or cognitive disorders, or participation in another conflicting clinical trial.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1600 (Estimated)
Dates: Start 2026-03-01 (Estimated); Primary Completion 2027-07-01 (Estimated); Study Completion 2027-08-01 (Estimated)

PRIMARY OUTCOMES:
Incidence of composite perioperative complications | From anesthesia induction up to 30 days after surgery
  This primary outcome measures the incidence of a composite of postoperative pulmonary complications (PPCs) within 30 days after surgery. The composite endpoint includes the occurrence of any one of the following predefined complications: pneumonia, respiratory failure, atelectasis requiring bronchoscopy, acute lung injury (ALI)/acute respiratory distress syndrome (ARDS), pulmonary embolism, bronchopleural fistula, pleural effusion requiring drainage, or pneumothorax requiring intervention. The assessment period begins at anesthesia induction and concludes 30 days post-surgery.
Postoperative recovery quality assessed by the QoR-15 score | At 24 hours after surgery
  This primary outcome measures the quality of patient recovery at 24 hours after surgery using the validated Quality of Recovery-15 (QoR-15) questionnaire. The QoR-15 score encompasses 15 items across five dimensions: physical comfort (5 items), emotional state (4 items), physical independence (2 items), psychological support (2 items), and pain (2 items). Each item is scored on a scale from 0 to 10. The total score ranges from 0 (extremely poor quality of recovery) to 150 (excellent quality of recovery). A higher total score indicates a better postoperative recovery experience from the patient's perspective.

SECONDARY OUTCOMES:
Length of postoperative hospital stay | From the day of surgery until the day of discharge, assessed up to 30 days.
  The duration of hospitalization in days, calculated from the day of surgery to the day of meeting discharge criteria (e.g., adequate pain control with oral analgesics, no air leak, afebrile, able to ambulate independently).
Incidence of intraoperative conversion | During the surgical procedure (from anesthesia induction until skin closure).
  The rate of conversion from non-intubated anesthesia to conventional intubated general anesthesia due to unacceptable surgical conditions (e.g., poor lung collapse, diaphragmatic movement) or patient safety concerns (e.g., hypoxemia, hypercapnia, hemodynamic instability).

CONTACTS AND LOCATIONS:
Locations (1):
- The First Affiliated Hospital of GZMU, Guangzhou, China

IPD SHARING:
Plan to Share IPD: Yes
De-identified individual participant data (IPD) that underlie the results reported in the primary and secondary outcomes of this study will be shared. This includes demographic data, perioperative parameters, and all assessed outcome measures.
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: The IPD and supporting documents will become available 6 months after the publication of the primary study results (the main manuscript). The data will be accessible for a period of 5 years.
Access Criteria: Researchers who provide a methodologically sound proposal for use in achieving the goals of the approved proposal may request access. Proposals should be directed to the corresponding author via email. Data requestors will need to sign a data access/use agreement. The shared data will be available for analyses aimed at replicating the study results, conducting secondary analyses, or performing meta-analyses.

REFERENCES:
- [Result] Wen Y, Liang H, Qiu G, Liu Z, Liu J, Ying W, Liang W, He J. Non-intubated spontaneous ventilation in video-assisted thoracoscopic surgery: a meta-analysis. Eur J Cardiothorac Surg. 2020 Mar 1;57(3):428-437. doi: 10.1093/ejcts/ezz279. PMID 31725158
- [Result] Myles PS, Shulman MA, Reilly J, Kasza J, Romero L. Measurement of quality of recovery after surgery using the 15-item quality of recovery scale: a systematic review and meta-analysis. Br J Anaesth. 2022 Jun;128(6):1029-1039. doi: 10.1016/j.bja.2022.03.009. Epub 2022 Apr 14. PMID 35430086
- [Result] Liu J, Liang H, Cui F, Liu H, Zhu C, Liang W, He J; International Tubeless-Video-Assisted Thoracoscopic Surgery Collaboration. Spontaneous versus mechanical ventilation during video-assisted thoracoscopic surgery for spontaneous pneumothorax: A randomized trial. J Thorac Cardiovasc Surg. 2022 May;163(5):1702-1714.e7. doi: 10.1016/j.jtcvs.2021.01.093. Epub 2021 Feb 3. PMID 33785209
- [Result] Zhang Z, Feng H, Zhao H, Hu J, Liu L, Liu Y, Li X, Xu L, Li Y, Lu X, Fu X, Yang H, Liu D. Sublobar resection is associated with better perioperative outcomes in elderly patients with clinical stage I non-small cell lung cancer: a multicenter retrospective cohort study. J Thorac Dis. 2019 May;11(5):1838-1848. doi: 10.21037/jtd.2019.05.20. PMID 31285876